CLINICAL TRIAL: NCT04278989
Title: Inhibition of Oral Tumorigenesis by Antitumor B
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Stuart Wong, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037907
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Cancer of the Oral Cavity
MeSH Terms: interventions — antitumor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-tumor B (Experimental): 1,200 mg three times a day.
  Interventions: Drug: Anti-tumor B

INTERVENTIONS:
Drug: Anti-tumor B — 1,200 mg, three times a day for seven to 28 days (dependent on scheduled surgery).
  Other Names: Zeng-Sheng-Ping; ACAPHA; ATB

SUMMARY:
This is a window of opportunity study of Anti-tumor B (ATB). Anti-tumor B is a botanical agent composed of six Chinese herbs: Sophora tonkinensis, Polygonum bistorta, Prunella vulgaris, Sonchus brachyotus, Dictamnus dasycarpus, and Dioscorea bulbifera.

DETAILED DESCRIPTION:
Upon initiating study treatment, patients will start taking the study drug. The duration of treatment will depend upon scheduling of their surgery--typically from the time surgery is scheduled it will be seven to 28 days. Four (300 mg) pills will be taken three times per day until the evening prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. In the event that the diagnosis of squamous cell cancer is made by an outside pathologist, hence not verified, the patient can start study agent administration but histological confirmation of squamous cell cancer (SCC) of the oral cavity (or histologic variants of SCC) by the pathologist must happen within seven days of registration in order to continue protocol therapy. Note: patients whose confirmatory biopsy fails to demonstrate invasive carcinoma will be excluded from continued participation in the study and considered a screen failure.
3. Clinical stage II-IVA (as defined by the American Joint Committee on Cancer (AJCC), 8th Edition), and amenable to surgical resection.
4. New diagnosis of oral SCC, new second primary, or recurrent oral SCC following a minimum remission of six months following previous definite surgery.
5. History and physical examination by an otolaryngologist and medical oncologist within 14 calendar days of study registration.
6. Zubrod/ECOG Performance status < 2.
7. Age ≥ 18 years.
8. Complete Blood Count (CBC)/differential obtained within 14 calendar days prior to registration, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3;
   * Platelets ≥ 100,000 cells/mm^3;
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable).
9. Adequate renal and hepatic function within 14 calendar days prior to registration, defined as follows:

   * Serum creatinine < 1.5 mg/dl or creatinine clearance (CCr) ≥ 50 ml/min within 14 calendar days prior to registration, determined by 24-hour collection or estimated by Cockcroft-Gault formula:
   * CCr male = [(140 - age) x (wt in kg)]
   * [(Serum Cr mg/dl) x (72)]
   * CCr female = 0.85 x (CrCl male)
10. Total bilirubin < 2 x the institutional upper limit of normal (ULN);
11. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x the institutional ULN;
12. Magnesium, calcium, glucose, potassium, and sodium within 14 calendar days prior to registration, with the following required parameters:

    * Magnesium: > 0.9 mg/dl or < 3 mg/dl;
    * Calcium: > 7 mg/dl or < 12.5 mg/dl;
    * Glucose: > 40 mg/dl or < 250 mg/dl;
    * Potassium: > 3 mmol/L or < 6 mmol/L;
    * Sodium: > 130 mmol/L or < 155 mmol/L.
13. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
14. Female subjects must meet one of the following:

    * Postmenopausal for at least one year before enrollment, OR
    * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
    * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agrees to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21days after the last dose of study agent, OR
    * Agrees to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
15. Male subjects, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

    * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
16. Enrollment on an interventional postoperative study is allowed if study agents do not overlap.
17. Gastric tube drug administration is permissible.

Exclusion Criteria:

1. Pregnant or lactating women are ineligible due to unforeseeable risks to embryo or fetus.
2. Concurrent use of any medicinal botanical, natural, or other herbal compounds.
3. Planned subtotal or debulking surgery is not permissible.
4. Prior systemic chemotherapy for oral SCC; note that prior chemotherapy for a different cancer is allowable.
5. Prior radiotherapy for oral SCC is permissible if disease free for one year since prior oral cancer treatment and free of significant late radiation effects.
6. Severe active comorbidity, such as uncontrolled cardiac disease, infection, and severe chronic obstructive pulmonary disease (COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Percent of Ki-67 positive cells | Baseline and after surgery (seven to 28 days after baseline)
  This measure is the immunohistochemical evaluation using the antihuman Ki-67 monoclonal antibody MIB-1 and reporting the percentage of positively stained malignant cells.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Wong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No